CLINICAL TRIAL: NCT00832910
Title: Body Image in Patients With Rheumatoid Arthritis
Brief Title: Assessment of Body Image in Patients With Rheumatoid Arthritis
Acronym: BIRA
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Renata Trajano Borges e Jorge, Federal University of São Paulo
Other Study IDs: FDAAA
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Body Image; Rheumatoid Arthritis
Keywords: Body image; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: None Retained — None Retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rheumatoid Arthritis group1: This group had patients with rheumatoid arthritis
- 2

SUMMARY:
Investigate body image of patients with rheumatoid arthritis, correlating with self-esteem, function and quality of life.

DETAILED DESCRIPTION:
Methods: Forty-three RA patients and thirty-nine control patients between 18 and 70 years were evaluated. The RA group was made up of individuals with a diagnosis of RA and the control group was made up of individuals from the community, paired for gender, age and body mass index. The patients were assessed with regard to body image (Body dysmorphic disorder examination (BDDE)), self-esteem (Rosenberg self-esteem scale), function (Health assessment questionnaire (HAQ)) and quality of life (Short form-36 (SF-36)).

ELIGIBILITY:
Inclusion Criteria:

* The RA group included patients between 18 and 70 years of age, of either gender, with an established diagnosis of RA based ACR criteria and belonging to functional classes I, II and III. The control group was made up of individuals from the community paired for gender, age and body mass index with RA group.

Exclusion Criteria:

* Individuals with fibromyalgia, neurological disease, psychiatric disorders or other severe co-morbidity were excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Rheumatoid arthritis in study group
  * Community sample in control group
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2007-06; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Body Dysmorphic Disorder Examination | baseline

SECONDARY OUTCOMES:
Short Form - 36 | baseline
Health assessment questionnaire | baseline
Rosenberg self-esteem scale | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Natour, Professor, Study Director — Federal University of São Paulo